CLINICAL TRIAL: NCT02106819
Title: Disorders of Emotional Communication in Patient With Cerebellar Dysfunction
Brief Title: Emotional Communication Disorders in Cerebellar Disease
Status: Completed | Type: Observational
Sponsor: University of Florida (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Other Study IDs: IRB201300595; 1R21AG044449-01A1 (NIH)
Record Dates: First submitted 2014-04-03; First posted 2014-04-08 (Estimated); Last update posted 2017-01-31 (Estimated); Status verified 2017-01

CONDITIONS: Cerebellar Diseases
Keywords: Cerebellar Ataxia; Emotions; Affective Prosody; Facial Expression; Magnetic Resonance Imaging
MeSH Terms: conditions — Cerebellar Diseases; Cerebellar Ataxia; Facial Expression | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Cerebellar Ataxia subjects: 40 individuals with either hereditary or sporadic ataxia will have testing of emotional communication ability and may have magnetic resonance imaging (MRI) of the brain.
  Interventions: Behavioral: Testing of emotional communication ability; Procedure: magnetic resonance imaging (MRI) of the brain
- Healthy Control subjects: 40 age matched controls will have testing of emotional communication ability and may have magnetic resonance imaging (MRI) of the brain.
  Interventions: Behavioral: Testing of emotional communication ability; Procedure: magnetic resonance imaging (MRI) of the brain

INTERVENTIONS:
Behavioral: Testing of emotional communication ability — Assessment of comprehension and expression of emotional facial and prosodic expressions and assessment of emotional reactivity via ratings of emotionally evocative pictures and words.
Procedure: magnetic resonance imaging (MRI) of the brain — Cerebellar participants who score at least 1 and a 1/2 standard deviations below the mean on the Florida Affect Battery and who have no contra-indications to scanning will be given an MRI. Healthy control participants who are willing and able to be scanned will also be given an MRI of the brain to use for analysis comparison.

SUMMARY:
The cerebellum has been linked to cognitive and emotional functions and there is increasing evidence that damage to posterior portions of the cerebellum can result in frontal-executive, visuospatial, and verbal deficits, including dysprosodia, and affective changes including blunting of affect or disinhibited and inappropriate behavior. Based on preliminary clinical observations and tests performed in the investigator's clinic, disorders of emotional communication may also be associated with cerebellar dysfunction. Emotional communication includes the production and comprehension of facial and prosodic expressions and is critical to maintaining positive and supportive relationships. Deficits in emotional communication can have devastating effects on relationships and on quality of life for those affected. Although deficits in affect and prosody have been reported in association with posterior cerebellar disorders, there are currently no studies systematically investigating emotional communication in individuals with cerebellar dysfunction. It is known that the cerebellum has strong connections with the cerebral cortex, especially the frontal lobes, and that cortical damage from stroke or neurodegenerative disease can result in disorders of emotional communication. Impairments in the integrity of cerebellar-cerebral networks from cerebellar disease may produce similar deficits in emotional communication. The purpose of this study is to systematically investigate and describe deficits in emotional communication in a series of patients with cerebellar disease. Participants will be individuals diagnosed with posterior cerebellar degeneration or damage from a non-hemorrhagic infarction, and age-matched neurologically healthy controls. Assessment will include a battery of tests of neuropsychological function as well as tests of emotional communication. Comprehension of emotional facial and prosodic expressions will be assessed as well as production of emotional communication. The expected outcomes will be to identify and describe deficits in production and comprehension of emotional prosodic and facial expressions and to describe the relationship between deficits in emotional communication and cerebellar atrophy with magnetic resonance imaging imaging (MRI) using voxel based morphometry (VBM).

DETAILED DESCRIPTION:
The specific aims of this proposal will investigate the hypothesis that cerebellar damage is associated with emotional communication deficits.

* Determine whether posterior cerebellar damage results in deficits in the production or comprehension of emotional facial expressions and/or vocal prosodic expressions
* Determine whether posterior cerebellar damage results in alterations in intensity of reaction to emotionally evocative pictures or emotionally evocative words
* Investigate the relationship between performance on tests of emotional communication and left versus right cerebellar atrophy with magnetic resonance imaging imaging (MRI) using voxel based morphometry (VBM) analysis

All subjects (cerebellar and control) will be given the following testing in a single session of lasting 3 to 3 and a half hours. Included will be tests to assess reading ability, naming ability, several tests of memory, a test of ability to discriminate between faces, tests of mental flexibility, and standardized questionnaires for depression, anxiety and emotional empathy. The tests include:

1. Wechsler Test of Adult Reading
2. Montreal Cognitive Assessment
3. Beck Depression Inventory - 2
4. Wisconsin Card Sorting test
5. Toronto Alexithymia Scale
6. Multi-Dimensional Emotional Empathy Scale

All subjects will also be given tests assessing emotional communication ability. Tests of recognition and expression of emotional tones of voice and facial expression will be performed. Expression of facial expressions and tones of voice will be video recorded so that blinded raters can compare the accuracy and intensity of facial expressions and tones of voice between the participants. Training for the raters will include familiarization with the descriptions of features for each emotion with respect to changes in pitch, loudness, and rate for prosody and changes in facial features for facial expression. Both intra- and inter-judge reliability will be calculated for these blinded judges. To supplement this perceptual analysis, the participant's responses will be recorded using VisiPitch IV software, a clinical instrument that performs sound analyses and calculates the variation in the range of fundamental frequency (i.e., pitch variation) across each sentence. The ability to manipulate pitch to produce varying prosodic contours is the most salient acoustical feature of affective prosody.

We will also assess intensity ratings and descriptions of emotional pictures and words using materials that have established rating norms. Participants will be shown a series of pictures and asked to rate the emotional intensity of the picture. They will also be asked to give a brief description of the picture. They will then be given a list of words, one at a time, and asked to rate the emotional intensity of these words.

Some of the cerebellar participants will also be asked to participate in a magnetic resonance imaging (MRI) scan of the brain if the testing listed above shows deficits in understanding or producing emotional facial expressions or tones of voice and if there are no reasons that would prevent them from being able to enter a scanner (determined by a standard MRI screen form). Healthy control participants may also be asked to participate in a magnetic resonance imaging (MRI) scan of the brain and if there are no reasons that would prevent them from being able to enter a scanner. The imaging data will be used to investigate if there is a relationship between our experimental subjects' performance on tests of emotional expression and left versus right cerebellar atrophy-injury in the cerebellar lobules with MRI imaging using a voxel based morphometry (VBM) approach. The same data from controls will be used for comparison. Neuroimaging data collection will be done using a Philips Achieva 3T scanner (Amsterdam, Netherlands) and a 32-channel SENSE head coil. Imaging collected will include anatomical T1-weighted imaging scans. Structural MP-RAGE T1-weighted scans will be acquired with 130-1.0 mm sagittal slices, FOV=240 mm (AP)-180 mm (FH), matrix= 256-192, TR= 9.90 ms, TE= 4.60 ms, Flip Angle= 8, voxel size= 1.0x 0.94x 0.94 mm. Structural data will be analyzed with FSL-VBM, an optimized VBM protocol carried out with FSL tools. First, structural images will be brain-extracted and grey matter-segmented before being registered to the MNI 152 standard space using non-linear registration The resulting images will be averaged and flipped along the x-axis to create a left-right symmetric, study-specific grey matter template. Second, all native grey matter images will be non-linearly registered to this study-specific template and "modulated" to correct for local expansion (or contraction) due to the non-linear component of the spatial transformation. The modulated grey matter images were then smoothed with an isotropic Gaussian kernel with a sigma of 6 mm. Finally, voxelwise GLM will be applied using permutation-based non-parametric testing, correcting for multiple comparisons across space.

ELIGIBILITY:
Inclusion Criteria:

* Men and women over the age of 18
* Individuals with cerebellar ataxia

Exclusion Criteria:

* Neurological signs reflecting major pathology in extrapyramidal, brainstem, cortical and visual systems
* Symptomatic cerebellar ataxia from alcohol, toxins, vitamin deficiency, and paraneoplastic cerebellar degeneration
* Dementia
* Current symptoms of depression or severe anxiety
* Currently on any psychotropic medication other than anti-depressants or history of a psychosis
* Severe impairments of hearing or vision
* Reading level less than 10th grade and/or history of learning disability
* Chronic medical and neurological diseases other than cerebellar (e.g., cardiac failure, renal disease, hepatic failure, stroke)
* History of severe head trauma (e.g., coma for more than one hour)

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The ataxia subjects will be recruited from the University of Florida Medical Center. The age matched controls have all been recruited and tested at this point.
Sampling Method: Non-Probability Sample
Enrollment: 56 (Actual)
Dates: Start 2014-04; Primary Completion 2016-12-31 (Actual); Study Completion 2016-12-31 (Actual)

PRIMARY OUTCOMES:
Florida Affect Battery | baseline
  Comprehension of emotional facial and prosodic expressions assessed via identification, discrimination and matching tasks.

SECONDARY OUTCOMES:
Perceptual rating of emotional expression | baseline
  Ability to express emotions by alterations of facial postures and changes in vocal prosody will be assessed imitatively and to-command. The expressions will be recorded and independently rated by three trained judges who will rate the type of facial or prosodic expression and the intensity (0-4).
Intensity and valence ratings of emotionally evocative pictures and words | baseline
  Comparison of participant ratings of valence and emotional intensity of words and pictures using items from a database of stimuli with normative ratings for emotional valence and arousal/intensity.
Magnetic resonance imaging of the brain | approximately one week post baseline
  Neuroimaging data collection will be done using a Philips Achieva 3T scanner (Amsterdam, Netherlands) and a 32-channel SENSE head coil. Imaging collected will include anatomical T1-weighted imaging scans.

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth M Heilman, MD, Principal Investigator — University of Florida
Locations (1):
- Department of Neurology, College of Medicine, University of Florida, Gainesville, Florida, United States

REFERENCES:
- [Background] Heilman KM, Leon SA, Burtis DB, Ashizawa T, Subramony SH. Affective communication deficits associated with cerebellar degeneration. Neurocase. 2014;20(1):18-26. doi: 10.1080/13554794.2012.713496. Epub 2012 Sep 28. PMID 23020242